CLINICAL TRIAL: NCT01373320
Title: Faith Moves Mountains: A CBPR Appalachian Wellness & Cancer Prevention Program
Brief Title: Faith Moves Mountains: A Community Based Participatory Research (CBPR) Appalachian Wellness & Cancer Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nancy Schoenberg (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Nancy Schoenberg, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R24MD002757 (NIH); R24MD002757 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer; Cervical Cancer; Breast Cancer; Colorectal Cancer
Keywords: Smoking cessation; Cancer screening; Appalachia; Group-randomized trial; Faith-placed
MeSH Terms: conditions — Lung Neoplasms; Uterine Cervical Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): Participants in this group are nested in churches which were randomly assigned to the treatment group.
  Interventions: Behavioral: Lay health advisor interactions
- Delayed Intervention (No Intervention): Participants in this group are nested in churches which were randomly assigned to the wait-list control group. They receive an educational luncheon focused on stress reduction during the intervention window for the Early Intervention group, and subsequently receive the intervention(s) for their selected target health behaviors at a later date.

INTERVENTIONS:
Behavioral: Lay health advisor interactions — For smoking cessation: Cooper-Clayton group sessions plus motivational interviewing, both delivered by local lay health advisor.
  For all cancer screenings: lay health advisor home visits incorporating motivational interviewing and focused on decreasing participant-identified barriers to screening.
  Arms: Early Intervention

SUMMARY:
The study purpose is to evaluate the effectiveness of a set of culturally appropriate, faith-placed lay health advisor interventions aimed at facilitating smoking cessation and increasing cancer screening among Appalachian participants.

DETAILED DESCRIPTION:
The developmental phase of this project incorporated community based participatory research (CBPR) principles to identify the needs and preferences of community members with regard to cancer prevention. In the intervention phase, this group-randomized trial administers and evaluates a set of culturally appropriate interventions aimed at facilitating smoking cessation and increasing cancer screening among participants in 6 distressed Appalachian counties. Faith institutions are recruited and randomized to treatment or wait-list control conditions, and participants are recruited and enrolled within those institutions. Participants select one or more targeted health behaviors from a menu including smoking cessation, colorectal cancer screening, cervical cancer screening, and breast cancer screening, and subsequently receive the intervention(s) aimed at their selected health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* For smoking cessation: age 18 or older; current cigarette smoker; able to provide informed consent
* For cervical cancer screening: female; age 18 or older AND outside of screening guidelines; able to provide informed consent
* For breast cancer screening: female; age 40 or older AND outside of screening guidelines; able to provide informed consent
* For colorectal cancer screening: age 40 or older AND outside of screening guidelines; able to provide informed consent

Exclusion Criteria:

* For smoking cessation: None
* For cervical cancer screening: History of cervical cancer; history of hysterectomy
* For breast cancer screening: History of breast cancer
* For colorectal cancer screening: History of colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants reporting the health behavior of interest (depending on which intervention component(s) were selected) | Assessed approximately 4 months after baseline
  For smoking cessation: Self-reported smoking status. For cancer screenings: Self-reported receipt of cervical, breast, and/or colorectal cancer screening. This assessment occurs after the Early Treatment group has completed the intervention.

SECONDARY OUTCOMES:
Change in stage of readiness to change the selected health behavior(s) from baseline | Assessed approximately 4 months after baseline
  Measured using reliable and valid instruments which were pretested in focus groups comprised of members of the target population. Positive change (i.e., increasing stage of readiness) from baseline to post-test will be coded as "1," while negative or no change will be coded "0." This assessment occurs after the Early Treatment group has completed the intervention.
Number of visits completed | Approximately 4 months after baseline
  This process measure will reflect the number of visits/classes attended by participants, as a means of assessing participation rate and feasibility.
Retention (i.e., number of participants who complete all planned assessment timepoints) | Approximately one year after baseline
  Retention numbers will be assessed as a process measure outcome. Participants who complete all study assessment timepoints will be coded as "1," while participants who drop out will be coded "0." Number/percentage of participants who remained enrolled and complete all study procedures and assessments will be used as an indicator of feasibility in the community setting.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenberg, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Faith Moves Mountains, Whitesburg, Kentucky, United States